CLINICAL TRIAL: NCT02964338
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group Study Comparing the Efficacy and Safety of 2 Dose Regimens (Intravenous/Subcutaneous and Subcutaneous) of TEV-48125 Versus Placebo for the Prevention of Chronic Cluster Headache
Brief Title: A Study Comparing the Efficacy and Safety of Fremanezumab (TEV-48125) for the Prevention of Chronic Cluster Headache (CCH)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility analysis revealed that the primary endpoint is unlikely to be met. There were no safety concerns observed with fremanezumab treatment in the trial.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30057; 2016-003171-21 (EudraCT Number)
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo via an approximately 1-hour intravenous infusion and as 3 subcutaneous injections at Week 0 followed by placebo administered as single subcutaneous injections at Weeks 4 and 8.
  Interventions: Drug: Placebo
- Fremanezumab 675/225/225 mg (Experimental): Participants received placebo via an approximately 1-hour intravenous infusion and fremanezumab at 675 milligrams (mg) as 3 subcutaneous injections (225 mg/1.5 milliliters [mL]) at Week 0 followed by fremanezumab at 225 mg administered as single subcutaneous injections (225 mg/1.5 mL) at Weeks 4 and 8.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Fremanezumab 900/225/225 mg (Experimental): Participants received fremanezumab at 900 mg via an approximately 1-hour intravenous infusion and placebo administered as 3 subcutaneous injections at Week 0 followed by fremanezumab at 225 mg administered as single subcutaneous injections (225 mg/1.5 mL) at Weeks 4 and 8.
  Interventions: Drug: Fremanezumab; Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab will be administered as per the dose and schedule specified in the respective arms.
  Other Names: TEV-48125
  Arms: Fremanezumab 675/225/225 mg; Fremanezumab 900/225/225 mg
Drug: Placebo — Placebo matching to fremanezumab will be administered as per the schedule specified in the respective arms.

SUMMARY:
The purpose of the current study is to evaluate the efficacy and safety of Fremanezumab (TEV-48125), in the prevention of CCH in adult participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a history of CCH according to the International Classification of Headache Disorders - 3 beta criteria (Headache Classification Committee of the International Headache Society [IHS] 2013) for greater than or equal to (≥)12 months prior to screening.
* The participant has a total body weight of ≥45 kilograms (kg) (99 pounds [lbs]).
* The participant is in good health in the opinion of the Investigator.
* Women of childbearing potential (WOCBP) whose male partners are potentially fertile (that is, no vasectomy) must use highly effective birth control methods for the duration of the study.
* Men must be sterile, or if they are potentially fertile/reproductively competent (not surgically [for example, vasectomy] or congenitally sterile) and their female partners are of childbearing potential, must agree to use, together with their female partners, acceptable birth control.
* If a participant is receiving Botox, it should be in a stable dose regimen, which is considered as having ≥2 cycles of Botox prior to screening. The participant should not receive Botox during the run-in period up to the evaluation period (12 weeks) where the primary endpoint is evaluated.

  * Additional criteria apply, please contact the Investigator for more information.

Exclusion Criteria:

* The participant has used systemic steroids for any medical reason (including treatment of the current cluster headache (CH) cycle within less than or equal to (≤)7 days prior to screening. The participant has used an intervention/device (for example, scheduled nerve blocks) for headache during the 4 weeks prior to screening.
* The participant has clinically significant hematological, renal, endocrine, immunologic, pulmonary, gastrointestinal, genitourinary, cardiovascular, neurologic, hepatic, or ocular disease at the discretion of the Investigator.
* The participant has evidence or medical history of clinically significant psychiatric issues determined at the discretion of the Investigator.
* The participant has a past or current history of cancer or malignant tumor in the past 5 years, except for appropriately treated non-melanoma skin carcinoma.
* The participant is pregnant or lactating.
* The participant has a history of hypersensitivity reactions to injected proteins, including monoclonal antibodies.
* The participant has participated in a clinical study of a monoclonal antibody within 3 months or 5 half-lives before administration of the first dose of the investigational medicinal product (IMP), whichever is longer, unless it is known that the participant received placebo during the study.
* The participant has a history of prior exposure to a monoclonal antibody targeting the calcitonin gene-related peptide (CGRP) pathway (AMG 334, ALD304, LY2951742, or fremanezumab). If participant has participated in a clinical study with any of these monoclonal antibodies, it has to be confirmed that the participant received placebo in order to be eligible for this study.
* The participant is an employee of the sponsor/participating study center who is directly involved in the study or is the relative of such an employee.
* The participant has an active implant for neurostimulation used in the treatment of CH.
* The participant is a member of a vulnerable population (for example, people kept in detention).
* The participant has a history of alcohol abuse prior to screening and/or drug abuse that in the Investigator's opinion could interfere with the study evaluations or the participant's safety.

  * Additional criteria apply, please contact the Investigator for more information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (83):
- United States (32):
  - Teva Investigational Site 13834, Phoenix, Arizona
  - Teva Investigational Site 13819, Canoga Park, California
  - Teva Investigational Site 13811, Santa Monica, California
  - Teva Investigational Site 13823, Stanford, California
  - Teva Investigational Site 13837, Aurora, Colorado
  - Teva Investigational Site 13814, Colorado Springs, Colorado
  - Teva Investigational Site 13836, Denver, Colorado
  - Teva Investigational Site 13813, Englewood, Colorado
  - Teva Investigational Site 13821, New Haven, Connecticut
  - Teva Investigational Site 13812, Stamford, Connecticut
  - Teva Investigational Site 13810, Gainesville, Florida
  - Teva Investigational Site 13815, Orlando, Florida
  - Teva Investigational Site 13829, Ormond Beach, Florida
  - Teva Investigational Site 13830, St. Petersburg, Florida
  - Teva Investigational Site 13840, Tampa, Florida
  - Teva Investigational Site 34222, Augusta, Georgia
  - Teva Investigational Site 13833, Columbus, Georgia
  - Teva Investigational Site 13826, Chicago, Illinois
  - Teva Investigational Site 13818, Ann Arbor, Michigan
  - Teva Investigational Site 13835, Las Vegas, Nevada
  - Teva Investigational Site 13832, Las Vegas, Nevada
  - Teva Investigational Site 13831, Lebanon, New Hampshire
  - Teva Investigational Site 13820, Princeton, New Jersey
  - Teva Investigational Site 13827, Albuquerque, New Mexico
  - Teva Investigational Site 13816, Amherst, New York
  - Teva Investigational Site 13817, New York, New York
  - Teva Investigational Site 13809, Raleigh, North Carolina
  - Teva Investigational Site 13839, Salisbury, North Carolina
  - Teva Investigational Site 13825, Cleveland, Ohio
  - Teva Investigational Site 13824, Philadelphia, Pennsylvania
  - Teva Investigational Site 13841, Richmond, Texas
  - Teva Investigational Site 13822, Virginia Beach, Virginia
- Australia (5):
  - Teva Investigational Site 78120, Auchenflower
  - Teva Investigational Site 78118, Clayton
  - Teva Investigational Site 78123, Melbourne
  - Teva Investigational Site 78122, Parkville
  - Teva Investigational Site 78121, Randwick
- Canada (3):
  - Teva Investigational Site 11132, Newmarket, Ontario
  - Teva Investigational Site 11130, Calgary
  - Teva Investigational Site 11131, Toronto
- Finland (3):
  - Teva Investigational Site 40030, Helsinki
  - Teva Investigational Site 40031, Oulu
  - Teva Investigational Site 40029, Turku
- Germany (7):
  - Teva Investigational Site 32666, Berlin
  - Teva Investigational Site 32667, Bochum
  - Teva Investigational Site 32660, Essen
  - Teva Investigational Site 32665, Hamburg
  - Teva Investigational Site 32662, Kiel
  - Teva Investigational Site 32661, Königstein im Taunus
  - Teva Investigational Site 32663, Rostock
- Israel (8):
  - Teva Investigational Site 80124, Ashkelon
  - Teva Investigational Site 80122, Hadera
  - Teva Investigational Site 80125, Holon
  - Teva Investigational Site 80121, Jerusalem
  - Teva Investigational Site 80123, Netanya
  - Teva Investigational Site 80120, Ramat Gan
  - Teva Investigational Site 80127, Tel Aviv
  - Teva Investigational Site 80126, Tel Aviv
- Italy (6):
  - Teva Investigational Site 30190, Milan
  - Teva Investigational Site 30192, Modena
  - Teva Investigational Site 30194, Napoli
  - Teva Investigational Site 30193, Pavia
  - Teva Investigational Site 30191, Rome
  - Teva Investigational Site 30189, Rome
- Netherlands (3):
  - Teva Investigational Site 38118, Leiden
  - Teva Investigational Site 38119, Nijmegen
  - Teva Investigational Site 38117, Zwolle
- Poland (5):
  - Teva Investigational Site 53380, Bialystok
  - Teva Investigational Site 53383, Krakow
  - Teva Investigational Site 53379, Krakow
  - Teva Investigational Site 53382, Lodz
  - Teva Investigational Site 53381, Szczecin
- Spain (5):
  - Teva Investigational Site 31211, Galdakao
  - Teva Investigational Site 31214, Madrid
  - Teva Investigational Site 31213, Seville
  - Teva Investigational Site 31212, Valladolid
  - Teva Investigational Site 31215, Zaragoza
- Sweden (2):
  - Teva Investigational Site 42047, Huddinge
  - Teva Investigational Site 42045, Vällingby
- United Kingdom (4):
  - Teva Investigational Site 34224, Glasgow
  - Teva Investigational Site 34220, London
  - Teva Investigational Site 34223, London
  - Teva Investigational Site 34221, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a history of chronic cluster headache (CCH) were enrolled. Eligible participants entered baseline cluster headache (CH) attack information into an electronic diary device daily for greater than or equal to (≥)4 weeks during the Baseline Period.
Pre-assignment Details: A total of 259 participants were randomly assigned with stratification based on sex, country, and baseline concomitant preventive medication use (yes/no) to either placebo, fremanezumab 675/225/225 milligrams (mg), or fremanezumab 900/225/225 mg treatment groups in a 1:1:1 ratio.
Groups:
- Fremanezumab 675/225/225 mg: Participants received placebo via an approximately 1-hour intravenous infusion and fremanezumab at 675 mg as 3 subcutaneous injections (225 mg/1.5 milliliters [mL]) at Week 0 followed by fremanezumab at 225 mg administered as single subcutaneous injections (225 mg/1.5 mL) at Weeks 4 and 8.
Period: Overall Study
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Started (Intent-to-Treat (ITT) Analysis Set: All randomized participants) | 84 | 88 | 87
Safety Analysis Set (All randomized participants who received at least 1 dose of study drug.) | 83 | 88 | 87
Full Analysis Set (ITT analysis set, received ≥1 dose of study drug, ≥10 days of postbaseline efficacy assessments) | 81 | 86 | 87
Completed | 67 | 64 | 68
Not Completed | 17 | 24 | 19
Not completed — Sponsor terminated study for futility | 12 | 15 | 14
Not completed — Lack of Efficacy | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Non-compliant with e-diary | 0 | 1 | 0
Not completed — Did not meet criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set included all randomized participants.
Groups:
- Fremanezumab 675/225/225 mg: Participants received placebo via an approximately 1-hour intravenous infusion and fremanezumab at 675 mg as 3 subcutaneous injections (225 mg/1.5 mL) at Week 0 followed by fremanezumab at 225 mg administered as single subcutaneous injections (225 mg/1.5 mL) at Weeks 4 and 8.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg | Total
Number analyzed (Participants) | 84 | 88 | 87 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.29) | 45.3 (11.40) | 43.8 (12.92) | 45.1 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 36 | 107
  Male | 49 | 52 | 51 | 152
Race/Ethnicity, Customized [Number; unit: participants]
  White | 79 | 83 | 79 | 241
  Black or African American | 4 | 4 | 8 | 16
  Asian | 0 | 1 | 0 | 1
  American Indian or Alaska native | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Middle Eastern | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 77 | 78 | 83 | 238
  Hispanic or Latino | 5 | 9 | 4 | 18
  Missing Ethnicity | 2 | 1 | 0 | 3
Number of CH Attacks During the Baseline Period [Mean (Standard Deviation); unit: CH attacks] — CH attack defined as a severe/very severe unilateral orbital, supraorbital, and/or temporal pain lasting 15-180 minutes with either or both of following 2 categories: 1) ≥1 of following symptoms/signs, ipsilateral to headache: -conjunctival injection and/or lacrimation; -nasal congestion and/or rhinorrhea; -eyelid edema; -forehead and facial sweating; -forehead and facial flushing; -sensation of fullness in ear; -miosis and/or ptosis. 2) sense of restlessness or agitation. Baseline period (≥4 weeks) defined as date informed consent was signed up to day before first dose of study drug.
  CH attacks | 38.0 (33.88) | 33.9 (27.37) | 44.0 (43.78) | 38.6 (35.75)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Overall Monthly Average Number of CH Attacks Up to Week 12
Description: A CH attack was defined as a severe or very severe unilateral orbital, supraorbital, and/or temporal pain lasting 15 to 180 minutes with either or both of the following 2 categories: 1) at least 1 of the following symptoms or signs, ipsilateral to the headache: -conjunctival injection and/or lacrimation; -nasal congestion and/or rhinorrhea; -eyelid edema; -forehead and facial sweating; -forehead and facial flushing; -sensation of fullness in the ear; -miosis and/or ptosis. 2) a sense of restlessness or agitation. Least Squares (LS) mean calculated using analysis of covariance (ANCOVA) model with baseline preventive medication use (yes or no), sex, region (United States [US]/Canada or other), and treatment as fixed effects and the baseline number of CH attacks as a covariate. Change from baseline in the overall monthly average number of CH attacks during the 12-week period after administration of the first dose of study drug (based on Week 0 to 12 data) is reported.
Time Frame: Baseline Period (from at least Week -4 to Week 0), Up to Week 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had at least 10 days of postbaseline efficacy assessments by the Week 12 assessment.
Measure: Least Squares Mean (Standard Error); unit: CH attacks/month
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 81 | 86 | 87
CH attacks/month | -12.2 (2.32) | -8.7 (2.26) | -15.5 (2.24)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675/225/225 mg; Test type: Other; p = 0.2741, ANCOVA — Threshold for significance at 0.05 level; Least square (LS) mean difference = 3.5, 95% CI 2-sided [-2.80 to 9.82]
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 900/225/225 mg; Test type: Other; p = 0.3047, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -3.3, 95% CI 2-sided [-9.59 to 3.01]

2. Secondary Outcome: Percentage of Participants With a ≥50% Reduction From Baseline in the Monthly Average Number of CH Attacks Up to Week 12
Description: A CH attack was defined as a severe or very severe unilateral orbital, supraorbital, and/or temporal pain lasting 15 to 180 minutes with either or both of the following 2 categories: 1) at least 1 of the following symptoms or signs, ipsilateral to the headache: -conjunctival injection and/or lacrimation; -nasal congestion and/or rhinorrhea; -eyelid edema; -forehead and facial sweating; -forehead and facial flushing; -sensation of fullness in the ear; -miosis and/or ptosis. 2) a sense of restlessness or agitation.
Time Frame: Baseline Period (from at least Week -4 to Week 0) up to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 81 | 86 | 87
percentage of participants | 40 | 40 | 45

3. Secondary Outcome: Mean Change From Baseline in the Monthly Average Number of CH Attacks at Week 4 and Week 12
Description: A CH attack was defined as a severe or very severe unilateral orbital, supraorbital, and/or temporal pain lasting 15 to 180 minutes with either or both of the following 2 categories: 1) ≥1 of the following symptoms or signs, ipsilateral to the headache: -conjunctival injection and/or lacrimation; -nasal congestion and/or rhinorrhea; -eyelid edema; -forehead and facial sweating; -forehead and facial flushing; -sensation of fullness in the ear; -miosis and/or ptosis. 2) a sense of restlessness or agitation. Mean change from baseline in monthly average number of CH attacks during 4-week period after administration of first dose of study drug (based on Week 0 to 4 data) and during 4-week period after administration of third dose of study drug (based on Week 8 to 12 data) is reported.
Time Frame: Baseline Period (from at least Week -4 to Week 0), Week 4 and Week 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug and had at least 10 days of postbaseline efficacy assessments by the Week 12 assessment. Here, 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: CH attacks/month
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 81 | 86 | 87
CH attacks/month
  Change at Week 4 | -10.4 (17.22) | -7.7 (19.53) | -15.0 (24.17)
  Change at Week 12: number analyzed (Participants) | 67 | 62 | 72
  Change at Week 12 | -12.6 (25.72) | -3.1 (34.42) | -17.9 (25.98)

4. Secondary Outcome: Mean Change From Baseline in the Overall Weekly Average Number of Days With Use of Cluster-Specific Acute Headache Medications (Triptans and Ergot Compounds) Up to Week 12
Description: A maximum of 2 concomitant preventive medications for CH were allowed during the study. Participants must have been on a stable dose and regimen of the concomitant medication for at least 2 weeks before screening and throughout the study. Baseline data and the mean change from baseline in the overall weekly average number of days with the use of cluster-specific acute headache medications (triptans and ergot compounds) during the 12-week period after administration of the first dose of study drug (based on Week 0 to 12 data) is reported.
Time Frame: Baseline Period (from at least Week -4 to Week 0), Up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days of use/week
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 81 | 86 | 87
days of use/week
  Baseline | 2.4 (2.42) | 2.4 (2.18) | 2.2 (2.27)
  Change at Week 12 | -0.7 (1.34) | -0.8 (1.57) | -0.8 (1.20)

5. Secondary Outcome: Mean Change From Baseline in the Weekly Average Number of Days Oxygen Was Used to Treat CCH Up to Week 12
Description: Baseline data and the mean change from baseline in the overall weekly average number of days oxygen was used to treat CCH during the 12-week period after administration of the first dose of study drug (based on Week 0 to 12 data) is reported.
Time Frame: Baseline Period (from at least Week -4 to Week 0), Up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days of use/week
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 81 | 86 | 87
days of use/week
  Baseline | 2.2 (2.59) | 1.9 (2.53) | 1.9 (2.59)
  Change at Week 12 | -0.5 (1.35) | -0.5 (1.35) | -0.5 (1.09)

6. Secondary Outcome: Number of Participants Who Perceived Improvement of CH-Associated Pain From Baseline as Measured by the Patient-Perceived Satisfactory Improvement (PPSI) Scale at Weeks 1, 4, 8, and 12
Description: The PPSI assessment was developed to measure pain intensity and was adjusted for CH symptoms improvement. Participants marked the level of CH-associated pain and indicated if pain is "1=much worse," "2=moderately worse," "3=slightly worse," "4=unchanged," "5=slightly improved," "6=moderately improved," or "7=much improved" compared with 4 weeks prior. PPSI was defined as the change in pain that corresponds with a minimal rating of "5=slightly improved." Data at Week 1 was recorded on Day 7 in the electronic diary device at home. Week 12 data also included assessment at the early withdrawal visit for participants who discontinued the study early.
Time Frame: Baseline and Weeks 1, 4, 8, and 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 81 | 86 | 87
Participants
  Much worse, Baseline | 3 | 1 | 1
  Moderately worse, Baseline | 1 | 4 | 4
  Slightly worse, Baseline | 1 | 5 | 4
  Unchanged, Baseline | 69 | 72 | 75
  Slightly improved, Baseline | 5 | 3 | 3
  Moderately improved, Baseline | 1 | 1 | 0
  Much improved, Baseline | 1 | 0 | 0
  Missing, Baseline | 0 | 0 | 0
  Much worse, Week 1 | 0 | 3 | 3
  Moderately worse, Week 1 | 0 | 2 | 1
  Slightly worse, Week 1 | 0 | 2 | 5
  Unchanged, Week 1 | 35 | 31 | 26
  Slightly improved, Week 1 | 23 | 20 | 32
  Moderately improved, Week 1 | 5 | 4 | 8
  Much improved, Week 1 | 6 | 13 | 8
  Missing, Week 1 | 12 | 11 | 4
  Much worse, Week 4 | 0 | 1 | 0
  Moderately worse, Week 4 | 1 | 2 | 3
  Slightly worse, Week 4 | 1 | 2 | 2
  Unchanged, Week 4 | 24 | 24 | 25
  Slightly improved, Week 4 | 30 | 17 | 25
  Moderately improved, Week 4 | 5 | 9 | 12
  Much improved, Week 4 | 12 | 18 | 11
  Missing, Week 4 | 8 | 13 | 9
  Much worse, Week 8 | 3 | 2 | 0
  Moderately worse, Week 8 | 1 | 3 | 3
  Slightly worse, Week 8 | 3 | 4 | 5
  Unchanged, Week 8 | 27 | 18 | 24
  Slightly improved, Week 8 | 18 | 12 | 13
  Moderately improved, Week 8 | 10 | 13 | 14
  Much improved, Week 8 | 4 | 12 | 15
  Missing, Week 8 | 15 | 22 | 13
  Much worse, Week 12 | 0 | 2 | 1
  Moderately worse, Week 12 | 3 | 5 | 3
  Slightly worse, Week 12 | 4 | 6 | 6
  Unchanged, Week 12 | 29 | 27 | 31
  Slightly improved, Week 12 | 21 | 18 | 15
  Moderately improved, Week 12 | 8 | 11 | 11
  Much improved, Week 12 | 13 | 14 | 12
  Missing, Week 12 | 3 | 3 | 8

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the Investigator on a scale of mild, moderate and severe, with severe as an AE that prevents usual activities. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants
  Any AE | 43 | 51 | 49
  Severe AE | 3 | 1 | 3
  Treatment-related AE | 17 | 23 | 28
  Serious AE | 2 | 2 | 3
  AE leading to discontinuation | 2 | 1 | 2

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory (Serum Chemistry, Hematology, and Urinalysis) Abnormal Results
Description: Serum chemistry, hematology, urinalysis laboratory tests with potentially clinically significant abnormal findings included: Alanine Aminotransferase (units/liter [U/L]) ≥3*upper limit of normal (ULN); Aspartate Aminotransferase (U/L) ≥3*ULN; Bilirubin (Total) ≥34.2 micromole/liter (umol/L); Blood Urea Nitrogen ≥10.71 millimole (mmol)/L; Creatinine ≥177 umol/L; Gamma Glutamyl Transferase (U/L) ≥3*ULN; hemoglobin less than (<)115 grams (g)/L (males) or less than or equal to (≤)95 g/L (females); leukocytes ≥20*10^9/L or ≤3*10^9/L; Eosinophils/Leukocytes ≥10%; Hematocrit <0.37 L/L (males) and <0.32 L/L (females); platelets ≥700*10^9/L or ≤75*10^9/L; blood ≥2 unit increase from baseline; urine glucose (milligrams/decilitre [mg/dL]) ≥2 U increase from baseline; ketones (mg/dL) ≥2 U increase from baseline; urine protein (mg/dL) ≥2 U increase from baseline. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants
  With at least 1 serum chemistry abnormality | 1 | 2 | 0
  With at least 1 hematology abnormality | 2 | 1 | 3
  With at least 1 urinalysis abnormality | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Shift From Baseline to Endpoint in Coagulation Laboratory Test Results
Description: Coagulation parameters included: prothrombin time (PT) (seconds) and prothrombin international normalized ratio (INR). Shifts represented as Baseline - endpoint value (last observed post-baseline value). Shifts from baseline to endpoint were summarized using participant counts grouped into three categories: - Low (below normal range) - Normal (within the normal range of 9.4 to 12.5 seconds) - High (above normal range). Missing PT and prothrombin INR shift data are also presented. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Here, 'Number analyzed' signifies participants evaluable at the timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants
  PT: Low-Low | 0 | 0 | 0
  PT: Low-Normal | 0 | 0 | 0
  PT: Low-High | 0 | 0 | 0
  PT: Normal-Low | 0 | 0 | 0
  PT: Normal-Normal | 68 | 69 | 62
  PT: Normal-High | 3 | 2 | 5
  PT: High-Low | 0 | 0 | 0
  PT: High-Normal | 5 | 8 | 11
  PT: High-High | 5 | 4 | 3
  PT: Missing | 2 | 5 | 6
  Prothrombin INR: Low-Low | 0 | 0 | 0
  Prothrombin INR: Low-Normal | 0 | 0 | 0
  Prothrombin INR: Low-High | 0 | 0 | 0
  Prothrombin INR: Normal-Low | 0 | 0 | 0
  Prothrombin INR: Normal-Normal | 70 | 71 | 69
  Prothrombin INR: Normal-High | 4 | 2 | 5
  Prothrombin INR: High-Low | 0 | 0 | 0
  Prothrombin INR: High-Normal | 5 | 7 | 6
  Prothrombin INR: High-High | 2 | 3 | 1
  Prothrombin INR: Missing | 2 | 5 | 6

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Potentially clinically significant abnormal vital signs findings included: pulse rate ≤50 beats/minute (bpm) and decrease of ≥15 bpm, or ≥120 bpm and increase of ≥15 bpm; systolic blood pressure ≤90 millimeters of mercury (mmHg) and decrease of ≥20 mmHg, or ≥180 mmHg and increase of ≥20 mmHg; diastolic blood pressure ≤50 mmHg and decrease of ≥15 mmHg, or ≥105 mmHg and increase of ≥15 mmHg; respiratory rate <10 breaths/minute; and body temperature ≥38.3 degrees centigrade and change of ≥1.1 degrees centigrade. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants | 3 | 0 | 0

11. Secondary Outcome: Number of Participants With Shift From Baseline to Endpoint (Last Assessment) in Electrocardiogram (ECG) Parameters
Description: ECG parameters included: heart rate, PR interval, QRS interval, QT interval corrected using the Fridericia formula (QTcF), QT interval corrected using the Bazett's formula (QTcB) and RR interval. Shifts represented as Baseline - endpoint value (last observed post-baseline value). Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding. Missing ECG shift data are also presented. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline to Week 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants
  Normal / Normal | 47 | 46 | 45
  Normal / NCS | 8 | 11 | 14
  Normal / CS | 0 | 0 | 0
  NCS / Normal | 10 | 7 | 8
  NCS / NCS | 15 | 20 | 12
  NCS / CS | 0 | 0 | 0
  CS / Normal | 0 | 0 | 0
  CS / NCS | 0 | 0 | 0
  CS / CS | 0 | 0 | 0
  Missing | 3 | 4 | 8

12. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Number of participants who reported treatment-emergent injection site reactions are summarized. Preferred terms from Medical Dictionary for Regulatory Activities (MedDRA) version 18.1 were offered without a threshold applied. Injection site reactions included injection site erythema, induration, pain, haemorrhage, bruising, hypersensitivity, swelling, rash, and flushing. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants
  Injection site erythema | 3 | 7 | 5
  Injection site induration | 3 | 6 | 6
  Injection site pain | 6 | 5 | 2
  Injection site haemorrhage | 0 | 0 | 2
  Injection site bruising | 0 | 0 | 1
  Injection site hypersensitivity | 0 | 1 | 0
  Injection site swelling | 2 | 0 | 0
  Injection site rash | 1 | 0 | 0
  Injection site flushing | 0 | 1 | 0

13. Secondary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior as Assessed by the Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
Description: eC-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent.
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
Number analyzed (Participants) | 83 | 88 | 87
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Fremanezumab 675/225/225 mg | Fremanezumab 900/225/225 mg
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/88 | 0/87
Serious Adverse Events (participants affected / at risk) | 2/83 | 2/88 | 3/87
Other Adverse Events (participants affected / at risk) | 18/83 | 22/88 | 19/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=83) | Fremanezumab 675/225/225 mg (N=88) | Fremanezumab 900/225/225 mg (N=87)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=83) | Fremanezumab 675/225/225 mg (N=88) | Fremanezumab 900/225/225 mg (N=87)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 3 (4)
Injection site erythema (General disorders) | 3 (4) | 7 (15) | 5 (6)
Injection site induration (General disorders) | 3 (8) | 6 (12) | 6 (12)
Injection site pain (General disorders) | 6 (11) | 5 (9) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 6 (7) | 8 (9)

LIMITATIONS AND CAVEATS:
Futility analysis revealed that the primary endpoint is unlikely to be met. There were no safety concerns observed with fremanezumab treatment in the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02964338/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT02964338/SAP_001.pdf